CLINICAL TRIAL: NCT05601362
Title: Evaluation of a Therapeutic Mobile App for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003315
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Gamified Attention Bias Modification (Active Comparator): Digital therapeutic intervention based on Attention Bias Modification Training (ABMT) designed to decrease negative attention bias.
  Interventions: Device: Gamified Attention Bias Modification
- Gamified Placebo Training (Sham Comparator): Identical version of the gamified behavioral intervention without manipulation designed to decrease negative attention bias
  Interventions: Device: Gamified Placebo Training

INTERVENTIONS:
Device: Gamified Attention Bias Modification — Gamified computerized behavioral therapy with therapeutic intervention based on Attention Bias Modification Training (ABMT).
  Arms: Gamified Attention Bias Modification
Device: Gamified Placebo Training — Placebo version of Gamified Attention Bias Modification. (Identical version of the gamified behavioral intervention without manipulation designed to decrease negative attention bias).
  Arms: Gamified Placebo Training

SUMMARY:
The purpose of this study is a preliminary evaluation of a gamified attention bias modification training (GAMBT) for reducing symptoms of depression and rumination. Individuals with elevated symptoms of depression will use the digital intervention over the course of 4 weeks. They will complete a brief (~5 question) survey daily, as well as weekly assessments.

DETAILED DESCRIPTION:
This study aims to assess the feasibility and efficacy of the digital therapeutic attention bias modification (ABM) intervention that targets and reduces negative attention bias among adults with elevated symptoms of depression. Consistent with the experimental therapeutics approach ABM has been shown to both reduce negative attention bias and improve symptoms of depression. However, engagement with these tasks have been mixed, with some participants describing traditional ABM tasks as boring. This had led to the development of gamified versions of ABM with the intent to improve participant engagement. Nevertheless, there have been very few rigorous trials of ABM for depression, and no one to our knowledge has used ecological momentary assessment to tease apart the mechanisms by which ABM can lead to improvements in depression symptoms.

Participants will access the intervention on their mobile smart phone and complete treatment over a period of 4 weeks. Enrolled participants will be randomly assigned to one of two groups: Gamified attention bias modification training, or gamified placebo training. They will complete brief (~5 questions) daily surveys, as well as weekly remote assessments of attention bias and depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to provide informed consent;
* fluent in English;
* normal or corrected-to-normal vision
* moderate or greater depression symptoms (defined as greater than or equal to 10 on the PHQ-8);
* attention bias for negative stimuli (operationalized as greater than an average of 6500 ms of dwell time on sad faces in an attention bias task);
* stable psychiatric and neurological medication usage.
* access to a smartphone for downloading the app and a laptop or desktop computer to complete the weekly assessments

Exclusion Criteria:

* recent heavy alcohol use defined as a score of 2 or higher on the PDSQ
* past or present comorbidity of other serious mental illness (e.g., schizophrenia, substance use disorder, bipolar disorder, etc.)
* previous experience with gamified attention bias modification app

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 8 (PHQ-8) | Baseline to Treatment End (4 weeks)
  8-item self-report measure of depression symptom severity (Range: 0-24, higher scores indicate greater depression severity)

SECONDARY OUTCOMES:
Ruminative Response Scale - Brooding subscale (RRS-B) | Baseline to Treatment End (4 weeks)
  5-item self-report measure of rumination frequency (Range: 1-20, higher scores indicate more rumination)
Perseverative Thinking Questionnaire (PTQ) -"Difficult to Disengage from" subscale | Baseline to Treatment End (4 weeks)
  3-item self-report measure of rumination frequency (Range: 0-12, higher scores indicate more rumination)
Inventory of Depression and Anxiety Symptoms (IDAS) Dysphoria subscale | Baseline to Treatment End (4 weeks)
  10-item measure of dysphoria and depression symptoms (Range: 10-50, higher scores indicate greater dysphoria)

OTHER OUTCOMES:
Attention bias (mousetracking) | Weekly assessment over 4 weeks
  Change in scan time for viewing sad stimuli assessed via mousetracking
General Rumination | daily over 4 weeks
  Change in rumination (assessed via smartphone-delivered ecological momentary assessment items used in prior EMA research (Smith et al., 2021)). (Range: 4-20, higher scores indicate more rumination)

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Eileen McNamara, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon study completion.